CLINICAL TRIAL: NCT02258802
Title: A Psychoeducational Intervention Model in Nutrition to Improve Nutritional Status in a Pilot Low Resource Population in the City of Saltillo, Coahuila Mexico.
Brief Title: Pilot Psychoeducational Intervention Model to Improve Nutritional Status in Low Resource Settings
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Monterrey (Other)
Collaborators: FEMSA Foundation (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 102014-CIE
Record Dates: First submitted 2014-09-30; First posted 2014-10-07 (Estimated); Last update posted 2016-05-13 (Estimated); Status verified 2016-05

CONDITIONS: Child Malnutrition; Child Overnutrition; Malnutrition in Children; Malnutrition, Child; Nutrition Disorders, Child; Malnutrition
Keywords: psychoeducational intervention; nutrition intervention; malnutrition; micronutrient deficiency; nutrition transition
MeSH Terms: conditions — Child Nutrition Disorders; Malnutrition | interventions — Nutritional Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Psychoeducational intervention (Experimental): Participants will be receiving a cooking lesson in their community every 2 weeks for 1 year.
  Interventions: Behavioral: Psychoeducational intervention
- Usual food practices (No Intervention): These are participants from the communities where the intervention is active but are not attending the cooking lessons.

INTERVENTIONS:
Behavioral: Psychoeducational intervention — A mobile kitchen visits the 5 selected communities every 2 weeks for a period of 1 year. A 30 minute cooking lesson is given by a trained instructor, the recipes have been designed to be quick and easy to make, use local and inexpensive ingredients, contain mostly vegetables and have a good taste. During the lesson, healthy habit and cooking tips are mentioned. A printed version of the recipe is given to every participant. Every lesson a different participant is encouraged to help prepare the recipe. At the end of the lesson all the participants get to taste the meal and express their opinion.
  Other Names: Psychoeducational intervention in nutrition
  Arms: Psychoeducational intervention

SUMMARY:
The purpose of this study is to develop, implement and evaluate a psychoeducational intervention focused to improve nutritional status, specifically micronutrients, of mothers and caregivers of children between the ages of 5 and 13 years and their children through providing healthy cooking lessons in their communities.

DETAILED DESCRIPTION:
Mexico's malnutrition problem goes beyond lack of food. Nutrition transition in our country has modified dietary patterns in a way that now we observe more and more a decrease in consumption of micronutrient rich foods, like vegetables, and an increase in consumption of high energy-dense foods with low content of micronutrients (highly processed foods). In Mexico, over 70% of the population presents an inadequate vegetable intake, with a higher prevalence in scholars (5 - 11 years), where only 17% of them consume >50% of the recommended vegetable intake. A vegetable poor diet is related to malnutrition, poor cognitive development and low physical performance. Added to this, Mexican families have lost the tradition of cooking at home. It is well known that different factors contribute to a population's diet and cooking at home as well as eating with the family have been identified as fundamental factors to promote a healthy diet. Therefore, the aim of this psychoeducational intervention in nutrition is to improve nutritional status in families, particularly mothers and caregivers of children between the ages of 5 and 13 years and their children through providing healthy cooking lessons in their communities where the optimal preparation and use of local foods based on vegetables is promoted at the same time the importance of cooking at home and eating as a family is highlighted.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 60 years
* Premenopausal
* BMI < 45 during enrollment
* Apparently healthy
* With a child in her care between the ages of 5 and 13 years

Exclusion Criteria:

* Pregnant or breastfeeding
* With a hysterectomy in the past 3 months
* Alcohol consumption > 14 drinks a week
* Use of vitamin supplements

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 65 (Actual)
Dates: Start 2014-06; Primary Completion 2015-07 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Change in food knowledge and behaviour | baseline, 6 months, 1 year
  questionnaire

SECONDARY OUTCOMES:
Change in vegetable intake | baseline, 1 year
  24 hour recall
Change in dietary practices | baseline, 6 months, 1 year
  questionnaire
Change in food waste | baseline, 6 months, 1 year
  questionnaire
Change in cognitive development in children | baseline, 1 year
  questionnaire
Change in anthropometry | baseline, 6 months, 1 year
  weight, height and waist circumference
Change in micronutrient status | baseline, 1 year
  serum sample
Change in inflammatory markers | baseline, 1 year
  serum sample

CONTACTS AND LOCATIONS:
Overall Officials: Ana Carla Cepeda-Lopez, PhD, Principal Investigator — Universidad de Monterrey

IPD SHARING:
Plan to Share IPD: No